CLINICAL TRIAL: NCT02542072
Title: Multi-Center Clinical Evaluation of Two Reusable Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: EX-MKTG-59 (VISA-406)
Record Dates: First submitted 2015-08-31; First posted 2015-09-04 (Estimated); Results first posted 2017-03-21 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- comfilcon A (Active Comparator): Participants were randomized to wear the comfilcon A lens pair for one month during the cross over study.
  Interventions: Device: comfilcon A
- samfilcon A (Active Comparator): Participants were randomized to wear the samfilcon A lens pair for one month during the cross over study.
  Interventions: Device: samfilcon A

INTERVENTIONS:
Device: comfilcon A — contact lens
  Arms: comfilcon A
Device: samfilcon A — contact lens
  Arms: samfilcon A

SUMMARY:
The purpose of this study is to compare the subjective performance of comfilcon A lens against samfilcon A lens after 4 weeks of reusable lens wear.

DETAILED DESCRIPTION:
This will be a 90 subject, randomized, bilateral, subject-masked, dispensing, cross-over study comparing comfilcon A versus samfilcon A lenses over 8 weeks of daily wear (2 x 4-weeks). Both eyes will wear the same lens (test or control) for 4 weeks in a randomized fashion. Subjects will be masked to lens type and investigators will be masked to the lens codes.

ELIGIBILITY:
Inclusion:

* Spherical distance Contact Lens prescription between -1.00 and -6.00D or +1.00 to +4.00D in both eyes (inclusive)
* Adapted soft Contact Lens wearers (i.e. >1 month), daily disposable and reusable lens wearers.
* Spectacle cylinder 0.75D in both eyes.
* Correctable to 6/9 (20/30) in both eyes
* Be between 18 and 50 years of age (inclusive)
* Able to read, comprehend and sign an informed consent
* Own a mobile phone and be willing to respond to Short Message Service (SMS) survey
* Willing to comply with the wear and study visit schedule

Exclusion:

* Existing Biofinity or Ultra wearers
* Any active corneal infection, injury or inflammation
* Systemic or ocular allergies, which might interfere with Contact Lens wear
* Systemic disease, which might interfere with Contact Lens wear
* Ocular disease, which might interfere with Contact Lens wear
* Strabismus or amblyopia
* Subjects who have undergone corneal refractive surgery
* Subjects with keratoconus or other severe corneal irregularity contraindicating lens wear
* Pregnant or lactating
* Use of systemic/topical medication contraindicating Contact Lens wear
* Diabetic
* Site employees or family members of site employees

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2015-08; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Young, Principal Investigator — VisionCare
Locations (5):
- United States (2):
  - Golden Optometric Group, Whittier, California
  - Complete Eye Care of Medina, Medina, Minnesota
- United Kingdom (3):
  - Brock & Houlford, Chew Magna, Bristol
  - Tempany's Boutique Opticians, Broadstone, Dorset
  - David Gould Opticians, Rawtenstall, Lancashire

RESULTS

PARTICIPANT FLOW:
Groups:
- Comfilcon A, Then Samfilcon A: Participants were randomized to wear the comfilcon A lens pair for one month, then cross over to the samfilcon A lens pair.
  comfilcon A: contact lens
  samfilcon A: contact lens
- Samfilcon A, Then Comfilcon A: Participants were randomized to wear the samfilcon A lens pair for one month then cross over to the comfilcon A lens pair.
  samfilcon A: contact lens
  comfilcon A: contact lens
Period: First Intervention (1 Month)
Arm/Group | Comfilcon A, Then Samfilcon A | Samfilcon A, Then Comfilcon A
Started | 44 | 46
Completed | 39 | 43
Not Completed | 5 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Lens discomfort | 1 | 2
Not completed — Protocol Violation | 1 | 0
Period: Second Intervention (1 Month)
Arm/Group | Comfilcon A, Then Samfilcon A | Samfilcon A, Then Comfilcon A
Started | 39 | 43
Completed | 37 | 43
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Lens discomfort | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Comfilcon A, Then Samfilcon A: Randomized participants who wore the comfilcon A lens pair for one month, then samfilcon A lens pair during the cross over study.
  comfilcon A: contact lenses
  samfilcon A: contact lenses
- Samfilcon A, Then Comfilcon A: Randomized participants who wore the samfilcon A lens pair for one month, then comfilcon A lens pair during the cross over study.
  comfilcon A: contact lenses
  samfilcon A: contact lenses
- Total: Total of all reporting groups
Arm/Group | Comfilcon A, Then Samfilcon A | Samfilcon A, Then Comfilcon A | Total
Number analyzed (Participants) | 44 | 46 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (9.3) | 30.8 (8.0) | 31.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 34 | 62
  Male | 16 | 12 | 28

OUTCOME MEASURES:

1. Primary Outcome: Comfort
Description: Subjective ratings of comfort (comfort after insertion, typical comfort just prior to removal, and overall comfort) for comfilcon A and samfilcon A assessed at baseline, 2 weeks, and 4 weeks. Scale of 0-10 (0=painful, 10=can't feel the lenses).
Time Frame: Baseline, 2 weeks, 4 weeks
Population: Number of participants analyzed is different from participant flow due to protocol deviations.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Habitual Lens (Baseline): Habitual data were collected of participants before lens dispensed.
- Comfilcon A (2 Weeks); Comfilcon A (4 Weeks): Participants were randomized to wear the comfilcon A lens pair for one month during the cross over study.
  comfilcon A: contact lens
- Samfilcon A (2 Weeks); Samfilcon A (4 Weeks): Participants were randomized to wear the samfilcon A lens pair for one month during the cross over study.
  samfilcon A: contact lens
Arm/Group | Habitual Lens (Baseline) | Comfilcon A (2 Weeks) | Samfilcon A (2 Weeks) | Comfilcon A (4 Weeks) | Samfilcon A (4 Weeks)
Number analyzed (Participants) | 90 | 82 | 82 | 82 | 80
units on a scale
  Comfort after insertion | 8.85 (1.92) | 9.06 (1.40) | 8.71 (1.81) | 8.84 (1.56) | 8.60 (1.80)
  Typical comfort just prior to removal | 7.72 (2.06) | 7.68 (2.11) | 7.09 (2.30) | 7.38 (2.32) | 6.94 (2.22)
  Overall comfort | 8.80 (1.75) | 8.33 (1.81) | 7.90 (1.90) | 8.01 (1.95) | 7.76 (1.76)

2. Secondary Outcome: Comfortable Wearing Time Via SMS (Short Message Service)
Description: Comfortable wearing times (WTs) via SMS (Short Message Service) for comfilcon A and samfilcon A lenses assessed at days 3, 12, and 26 at hours 8:00 am, 12:00 pm, 4:00 pm, and 8:00 pm. Scale of 0-10 (0=painful, 10=can't feel the lenses).
Time Frame: Days 3, 12, 26
Population: Number of participants analyzed may differ from participant flow due to protocol deviations.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Comfilcon A (Day 3); Comfilcon A (Day 12); Comfilcon A (Day 26): Participants were randomized to wear the comfilcon A lens pair for one month during the cross over study.
  comfilcon A: contact lens
- Samfilcon A (Day 3); Samfilcon A (Day 12); Samfilcon A (Day 26): Participants were randomized to wear the samfilcon A lens pair for one month during the cross over study.
  samfilcon A: contact lens
Arm/Group | Comfilcon A (Day 3) | Samfilcon A (Day 3) | Comfilcon A (Day 12) | Samfilcon A (Day 12) | Comfilcon A (Day 26) | Samfilcon A (Day 26)
Number analyzed (Participants) | 85 | 85 | 83 | 84 | 82 | 82
units on a scale
  8:00 am | 8.59 (1.85) | 8.82 (1.61) | 8.90 (1.46) | 8.84 (1.36) | 8.98 (1.45) | 8.51 (1.67)
  12:00 pm | 8.97 (1.26) | 9.07 (1.03) | 8.71 (1.87) | 8.55 (1.83) | 8.44 (1.74) | 8.11 (2.12)
  4:00 pm | 8.56 (1.80) | 8.65 (1.53) | 8.19 (1.84) | 8.03 (1.98) | 8.06 (1.85) | 8.07 (1.63)
  8:00 pm | 8.53 (1.52) | 8.30 (1.59) | 8.06 (1.93) | 7.84 (2.21) | 7.87 (2.25) | 7.82 (2.09)

3. Secondary Outcome: Wearing Times
Description: Average wear time and comfortable wearing times (WTs) in hours for habitual, comfilcon A, and samfilcon A lenses.
Time Frame: Baseline, 2 weeks, 4 weeks
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Habitual Lens (Baseline) | Comfilcon A (2 Weeks) | Samfilcon A (2 Weeks) | Comfilcon A (4 Weeks) | Samfilcon A (4 Weeks)
Number analyzed (Participants) | 90 | 82 | 82 | 82 | 80
hours
  Average wearing time | 6.16 (1.37) | 13.94 (1.82) | 13.68 (2.46) | 13.90 (2.18) | 13.93 (2.11)
  Comfortable wearing time | 12.79 (2.64) | 11.58 (3.05) | 11.28 (3.84) | 11.34 (3.48) | 11.02 (3.63)
  Maximum wearing time | 16.59 (2.90) | 16.15 (2.39) | 15.48 (2.48) | 16.04 (2.44) | 15.91 (2.35)

4. Secondary Outcome: Deterioration in Comfort
Description: Deterioration of comfortable wearing time for habitual, comfilcon A, samfilcon A lenses. Subjects answered 'yes' or 'no' to the following question 'does contact lens comfort deteriorate during wear?'. Yes=deterioration in comfort present, No=deterioration in comfort absent
Time Frame: Baseline, 2 weeks, 4 weeks
Measure: Number; unit: participants
Arm/Group | Habitual Lens (Baseline) | Comfilcon A (2 Weeks) | Samfilcon A (2 Weeks) | Comfilcon A (4 Weeks) | Samfilcon A (4 Weeks)
Number analyzed (Participants) | 90 | 82 | 82 | 82 | 80
participants
  Yes=deterioration in comfort present | 47 | 51 | 46 | 53 | 52
  No=deterioration in comfort absent | 43 | 31 | 36 | 29 | 28

5. Secondary Outcome: Vision Quality
Description: Vision quality of comfilcon A and samfilcon A lenses. Scale 0-10, 0=completely dissatisfied, 10=completely satisfied.
Time Frame: Baseline, 2 weeks, 4 weeks
Population: Number of participants analyzed differ from participant flow due to protocol deviations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Habitual Lens (Baseline) | Comfilcon A (2 Weeks) | Samfilcon A (2 Weeks) | Comfilcon A (4 Weeks) | Samfilcon A (4 Weeks)
Number analyzed (Participants) | 90 | 82 | 82 | 82 | 80
units on a scale | 9.31 (1.10) | 9.06 (1.15) | 8.49 (1.81) | 8.81 (1.55) | 8.34 (1.79)

6. Secondary Outcome: Overall Lens Handling
Description: Handling (ease of insertion and ease of removal) for comfilcon A and samfilcon A lenses. Scale 0-10, 0=very difficult to handle, 10=very easy to handle.
Time Frame: Baseline, 2 weeks, 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Habitual Lens (Baseline) | Comfilcon A (2 Weeks) | Samfilcon A (2 Weeks) | Comfilcon A (4 Weeks) | Samfilcon A (4 Weeks)
Number analyzed (Participants) | 90 | 82 | 82 | 82 | 80
units on a scale
  Ease of insertion | 9.31 (1.40) | 9.12 (1.56) | 8.96 (1.69) | 9.18 (1.48) | 8.83 (1.73)
  Ease of removal | 9.31 (1.38) | 8.94 (1.84) | 9.06 (1.53) | 8.86 (2.14) | 8.98 (1.48)

7. Secondary Outcome: Biomicroscopy Scores
Description: Biomicroscopy for comfilcon A and samfilcon A lens assessed. Scale 0-4 in 0.5 steps 0=none, 1=trace, 2=mild, 3=moderate, 4=severe
Time Frame: Baseline, 2 weeks, 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Groups:
- Habitual Lenses (Baseline): Habitual data were collected of participants before lens dispensed.
Arm/Group | Habitual Lenses (Baseline) | Comfilcon A (2 Weeks) | Samfilcon A (2 Weeks) | Comfilcon A (4 Weeks) | Samfilcon A (4 Weeks)
Number analyzed (Participants) | 90 | 82 | 82 | 82 | 80
Number analyzed (Eyes) | 180 | 164 | 164 | 164 | 160
units on a scale
  Limbal Hyperaemia | 0.39 (0.39) | 0.42 (0.50) | 0.45 (0.45) | 0.47 (0.48) | 0.49 (0.46)
  Bulbar Hyperaemia | 0.67 (0.53) | 0.60 (0.58) | 0.67 (0.57) | 0.61 (0.57) | 0.62 (0.52)
  Palpebral Conjunctiva | 0.53 (0.59) | 0.73 (0.75) | 0.72 (0.85) | 0.79 (0.77) | 0.78 (0.79)
  Corneal Staining | 0.39 (0.55) | 0.63 (0.66) | 0.56 (0.63) | 0.69 (0.70) | 0.56 (0.72)
  Conjunctival fluorescein staining | 0.67 (0.61) | 0.75 (0.66) | 1.23 (0.69) | 0.81 (0.67) | 1.19 (0.71)

8. Secondary Outcome: Lens Surface Wetting
Description: Lens surface wettability assessment for comfilcon A and samfilcon A lenses. Scale 0-4 in 0.5 steps, 0=very poor, 4=excellent
Time Frame: Baseline, 2 weeks, 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Groups:
- Comfilcon A (Baseline); Comfilcon A (2 Weeks); Comfilcon A (4 Weeks): Participants were randomized to wear the comfilcon A lens pair for one month during the cross over study.
  comfilcon A: contact lens
- Samfilcon A (Baseline); Samfilcon A (2 Weeks); Samfilcon A (4 Weeks): Participants were randomized to wear the samfilcon A lens pair for one month during the cross over study.
  samfilcon A: contact lens
Arm/Group | Comfilcon A (Baseline) | Samfilcon A (Baseline) | Comfilcon A (2 Weeks) | Samfilcon A (2 Weeks) | Comfilcon A (4 Weeks) | Samfilcon A (4 Weeks)
Number analyzed (Participants) | 87 | 85 | 82 | 82 | 82 | 80
Number analyzed (Eyes) | 174 | 170 | 164 | 164 | 164 | 160
units on a scale | 3.69 (0.51) | 3.61 (0.57) | 3.51 (0.56) | 3.37 (0.70) | 3.27 (0.85) | 3.22 (0.81)

9. Secondary Outcome: Film Deposits
Description: Front surface film deposits for comfilcon A and samfilcon A lenses. Scale 0-4, 0=No film, 1=Slight film visible only under magnification, 2=Moderate film only under magnification, 3=Moderate film visible to the naked eye, 4=Heavy film visible to the naked eye.
Time Frame: 2 weeks and 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Comfilcon A (2 Weeks) | Samfilcon A (2 Weeks) | Comfilcon A (4 Weeks) | Samfilcon A (4 Weeks)
Number analyzed (Participants) | 82 | 82 | 82 | 80
Number analyzed (Eyes) | 164 | 164 | 164 | 160
units on a scale | 0.12 (0.32) | 0.26 (0.63) | 0.35 (0.73) | 0.30 (0.63)

10. Secondary Outcome: White Spot Deposits
Description: Number of white spot deposits for comfilcon A and samfilcon A lenses.
Time Frame: 2 weeks and 4 weeks
Measure: Mean (Standard Deviation); unit: number of white spots
Units Other Than Participants: Eyes
Arm/Group | Comfilcon A (2 Weeks) | Samfilcon A (2 Weeks) | Comfilcon A (4 Weeks) | Samfilcon A (4 Weeks)
Number analyzed (Participants) | 82 | 82 | 82 | 80
Number analyzed (Eyes) | 164 | 164 | 164 | 160
number of white spots | 0.3 (1.0) | 0.4 (1.4) | 0.8 (2.6) | 0.7 (2.4)

11. Secondary Outcome: Visual Acuity (VA)
Description: Visual acuity (VA) for comfilcon A and samfilcon A lens wear is assessed using Snellen.
Time Frame: Baseline, 2 weeks, 4 weeks
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Habitual Lens (Baseline) | Comfilcon A (2 Weeks) | Samfilcon A (2 Weeks) | Comfilcon A (4 Weeks) | Samfilcon A (4 Weeks)
Number analyzed (Participants) | 90 | 82 | 82 | 82 | 80
LogMAR
  Distance Visual Acuity | -0.03 (0.08) | -0.04 (0.10) | -0.01 (0.10) | -0.03 (0.10) | -0.02 (0.12)
  Binocular Distance Visual Acuity | -0.07 (0.09) | -0.08 (0.10) | -0.07 (0.09) | -0.08 (0.10) | -0.07 (0.10)

12. Secondary Outcome: Lens Centration
Description: Lens centration will be recorded by degree and direction in the primary position. 0=Centered -optimal, 1=Decentered slightly, 2=Substantially decentered (>0.5mm)
Time Frame: Baseline, 2 weeks, 4 weeks
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Comfilcon A (Baseline) | Samfilcon A (Baseline) | Comfilcon A (2 Weeks) | Samfilcon A (2 Weeks) | Comfilcon A (4 Weeks) | Samfilcon A (4 Weeks)
Number analyzed (Participants) | 87 | 85 | 82 | 82 | 82 | 80
Number analyzed (Eyes) | 174 | 170 | 164 | 164 | 164 | 160
Eyes
  Centered - optimal | 173 | 153 | 162 | 152 | 163 | 156
  Decentered slightly | 1 | 16 | 2 | 12 | 1 | 4
  Substantially decentered | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Corneal Coverage
Description: Investigator assessment of corneal coverage for comfilcon A and samfilcon A lenes.
  Yes = coverage at all times or No = coverage incomplete
Time Frame: Baseline Visit, 2 weeks follow-up, 4-weeks follow-up
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Comfilcon A (Baseline) | Samfilcon A (Baseline) | Comfilcon A (2 Weeks) | Samfilcon A (2 Weeks) | Comfilcon A (4 Weeks) | Samfilcon A (4 Weeks)
Number analyzed (Participants) | 87 | 85 | 82 | 82 | 82 | 80
Number analyzed (Eyes) | 174 | 170 | 164 | 164 | 164 | 160
percentage of eyes
  Yes | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0
  No | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

14. Secondary Outcome: Post-Blink Movement
Description: Post-blink movement for comifilcon A and samfilcon A lenses are assessed. 0=Insufficient, unacceptable movement, 1=Minimal, but acceptable movement, 2=Optimal movement, 3=Moderate, but acceptable movement, 4=Excessive, unacceptable movement
Time Frame: Baseline, 2 weeks, 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Comfilcon A (Baseline) | Samfilcon A (Baseline) | Comfilcon A (2 Weeks) | Samfilcon A (2 Weeks) | Comfilcon A (4 Weeks) | Samfilcon A (4 Weeks)
Number analyzed (Participants) | 87 | 85 | 82 | 82 | 82 | 80
Number analyzed (Eyes) | 174 | 170 | 164 | 164 | 164 | 160
units on a scale | 1.91 (0.55) | 1.86 (0.58) | 1.84 (0.51) | 1.79 (0.58) | 1.87 (0.42) | 1.69 (0.50)

15. Secondary Outcome: Primary Gaze Lag
Description: Investigator assessment of primary gaze lag for comfilcon A and samfilcon A lenses. Scale 0-4, 0=Insufficient, unacceptable movement, 1=Minimal, but acceptable movement, 2=Optimal movement, 3=Moderate, but acceptable movement, 4=Excessive, unacceptable movement
Time Frame: Baseline, 2 weeks, and 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Comfilcon A (Baseline) | Samfilcon A (Baseline) | Comfilcon A (2 Weeks) | Samfilcon A (2 Weeks) | Comfilcon A (4 Weeks) | Samfilcon A (4 Weeks)
Number analyzed (Participants) | 87 | 85 | 82 | 82 | 82 | 80
Number analyzed (Eyes) | 174 | 170 | 164 | 164 | 164 | 160
units on a scale | 1.89 (0.55) | 1.82 (0.63) | 1.78 (0.54) | 1.69 (0.56) | 1.88 (0.48) | 1.71 (0.54)

16. Secondary Outcome: Lens Tightness Push-up
Description: Investigator assessment of lens tightness push-up for comfilcon A and samfilcon A lenses.
  Scale 0%-100% continuous scale, 100%=No movement, 50%=Optimum, 0%=Falls from cornea without lid support
Time Frame: Baseline, 2 weeks, 4 weeks
Measure: Mean (Standard Deviation); unit: percentage of mean lens tightness
Units Other Than Participants: Eyes
Arm/Group | Comfilcon A (Baseline) | Samfilcon A (Baseline) | Comfilcon A (2 Weeks) | Samfilcon A (2 Weeks) | Comfilcon A (4 Weeks) | Samfilcon A (4 Weeks)
Number analyzed (Participants) | 87 | 85 | 82 | 82 | 82 | 80
Number analyzed (Eyes) | 174 | 170 | 164 | 164 | 164 | 160
percentage of mean lens tightness | 48.9 (10.8) | 54.3 (11.9) | 50.6 (10.4) | 54.1 (9.9) | 50.3 (8.2) | 54.6 (8.4)

17. Secondary Outcome: Overall Fit Acceptance
Description: Overall fit acceptance for comfilcon A and samfilcon A lenses. Scale 0-4, 0=Should not be worn, 1=Borderline but unacceptable, 2=Minimum acceptable, early review, 3=Not perfect but okay to dispense, 4=Perfect
Time Frame: Baseline, 2 weeks, 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A (Baseline) | Samfilcon A (Baseline) | Comfilcon A (2 Weeks) | Samfilcon A (2 Weeks) | Comfilcon A (4 Weeks) | Samfilcon A (4 Weeks)
Number analyzed (Participants) | 87 | 85 | 82 | 82 | 82 | 80
units on a scale | 3.71 (0.45) | 3.63 (0.48) | 3.73 (0.44) | 3.63 (0.48) | 3.78 (0.42) | 3.66 (0.48)

18. Secondary Outcome: Dryness
Description: Subjective response of dryness for comfilcon A and samfilcon A lenses during a typical day of wear and prior to removal. Scale of 0-10, 10=No dryness, 0=Extremely dry
Time Frame: Baseline, 2 weeks, 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Habitual Lens (Baseline) | Comfilcon A (2 Weeks) | Samfilcon A (2 Weeks) | Comfilcon A (4 Weeks) | Samfilcon A (4 Weeks)
Number analyzed (Participants) | 90 | 82 | 82 | 82 | 80
units on a scale
  During a typical day of wear | 8.06 (2.24) | 7.98 (1.91) | 7.46 (2.12) | 7.71 (2.13) | 7.18 (2.22)
  Prior to removal | 7.57 (2.26) | 7.61 (2.12) | 6.83 (2.49) | 7.27 (2.49) | 6.60 (2.44)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the study duration (8 week wear period)
Description: Adverse events were assessed for during the study visits over the duration of the 8 week study.
Arm/Group | Comfilcon A | Samfilcon A
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/90
Other Adverse Events (participants affected / at risk) | 0/90 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other